CLINICAL TRIAL: NCT04601649
Title: Evaluating the Feasibility and Acceptability of "PrEP-Talk": A PrEP Uptake Intervention for Young Black MSM With Their Close Friends
Brief Title: PrEP Talk: PrEP Uptake With Young Black MSM and Their Close Friends
Acronym: PrEP-Talk
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California State University, Dominguez Hills (Other)
Responsible Party: Principal Investigator, Dr. Matt G. Mutchler, Principal Investigator, California State University, Dominguez Hills
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PrEP Talk with Friends
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: HIV Negative and Not Yet on PrEP

STUDY DESIGN:
Intervention Model Description: 30 friendship dyads (N=60) will be assigned to a control group and 30 friends dyads (N=60) will be assigned to the intervention group to collect feasibility and acceptability data.
Masking Description: None; this is a feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will take part in the PrEP Talk intervention sessions.
  Interventions: Behavioral: PrEP Talk
- Control (No Intervention): Participants will receive standard care.

INTERVENTIONS:
Behavioral: PrEP Talk — The study is designed to provide education, support, and referrals for PrEP.
  Arms: Intervention

SUMMARY:
Young Black MSM (YBMSM) are at critically high and disproportionate HIV risk. Reducing HIV incidence rates among YBMSM will likely require increased adoption of additional strategies such as pre-exposure prophylaxis (PrEP). PrEP is a FDA approved medication for HIV that also prevents HIV transmission when taken appropriately. Interventions are needed to address potential individual, social/cultural, and structural barriers to uptake and adherence of PrEP among YBMSM to help curb HIV infections. Our preliminary research suggests that some YBMSM feel concerned that PrEP is not effective or may be toxic, about being stigmatized for having HIV if they take PrEP, as well as concerns about access and side effects. For YBMSM, high levels of medical mistrust of HIV-related public health information and research may also be barriers. Therefore, we propose "PrEP-Talk", an intervention that will use a PrEP Counselor (PC) who can provide information and guidance to YBMSM as they weigh their options regarding HIV risk along with the inclusion of a close friend (CF) to support PrEP uptake and adherence. In order to address these critical and timely issues, we developed the following specific aims:

1. To develop and manualize "PrEP-Talk," which aims to increase PrEP uptake and adherence among YBMSM. This will be done through qualitative formative research (3 focus groups with 12-18 YBMSM and CF dyads, N=24-36); partnering with a community advisory board (comprised of individuals knowledgeable about HIV work with YBMSM); and field tests of the intervention with 5 YBMSM and CF dyads (N=10).
2. Examine feasibility, acceptability and indicators of preliminary efficacy of "PrEP-Talk" on PrEP uptake and adherence among YBMSM. This will be accomplished through a pilot randomized controlled trial (RCT) with 30 dyads (YBMSM and CFs) in the intervention and 30 YBMSM in the control (N=90). We will conduct assessments at baseline, 3-months and 6-months post-baseline. We will also assess PrEP uptake supportive communication at each intervention session and collect urine samples to measure a biomarker of PrEP uptake (initial adherence) from all YBMSM who report use of PrEP.

This proposed study is significant because our intervention may increase PrEP uptake and adherence, which may help to reduce HIV incidence among YBMSM. If the proposed intervention shows promise, we will prepare to undertake a full-scale R01-funded RCT.

DETAILED DESCRIPTION:
Young Black men who have sex with men (YBMSM) face a disproportionate burden of HIV infection. Pre-exposure prophylaxis (PrEP) is an effective tool for protecting individuals from HIV infection. However, uptake has been relatively slow among YBMSM (5-10%). 8 There is an urgent need to develop and test interventions to increase PrEP uptake with YBMSM, which is consistent with NIH priorities to examine the use of biomedical interventions for HIV prevention with high risk populations.

Our prior research indicates that many YBMSM are considering using PrEP, but they are skeptical about taking a pill daily for HIV prevention. 5 YBMSM's willingness to use PrEP is affected by many factors such as PrEP literacy, their own perceived low risk for HIV, concerns about taking the pill and side effects, medical mistrust, concerns about cost, lack of social support for using PrEP, and PrEP-related stigma. Consistent with our prior research showing the powerful influence of close social network members on HIV-related health behaviors, we have found that close friends of YBMSM can strongly influence YBMSM's' motivation to use PrEP via conversations with each other.

Guided by peer influence theory, a motivational interviewing (MI) approach and prior research, the goal of the proposed research is to develop, manualize, and evaluate a culturally-congruent intervention, "PrEP-Talk," which aims to increase PrEP uptake and adherence among YBMSM. We propose that their close friends can apply positive peer influence about taking PrEP. Our research is based on exploring how using MI with YBMSM and their close friends may help to overcome barriers to PrEP uptake and adherence.

We designed a dyad-level intervention concept for PrEP-Talk that involves three interconnected components to increase PrEP uptake: 1) a "PrEP Counselor" (PC), in which information and guidance will be provided to YBMSM and a Close Friend they select to help address barriers to making an informed decision regarding PrEP uptake, (2) a Close Friend (CF), defined as someone with whom the YBMSM has discussed sexual health topics in the past year (but not had sex with in the past year), who is aware that he has sex with men, and who agrees to support his PrEP uptake goals by engaging in dyad-level sessions about PrEP uptake and adherence with their friend, and (3) training on PrEP supportive communication (PSC) in every day conversations between YBMSM and CFs. PSC is talk between CFs that is well-informed and non-judgmental about PrEP, in which YBMSM discuss the pros and cons of PrEP use, helping YBMSM overcome barriers to uptake. All three components address the mechanisms of change (barriers and facilitators such as PrEP-related stigma, medical mistrust, concerns about cost, etc.) that are related to PrEP uptake and adherence among YBMSM. Culturally congruent referrals and linkages will also be provided. The proposed study is built on the scientific premise that peers, especially close friends, have a strong influence on health behaviors, through their communication about attitudes toward health topics such as PrEP uptake.

Our research has shown that YBMSM's CFs are particularly helpful in facilitating decisions about PrEP through providing supportive communication and that using MI can lead to increased antiretroviral therapy (ART) adherence among Black people living with HIV. 1, 4-7 In our proposed intervention, the PC will work with the YBMSM and the CF as they grapple with concerns about PrEP before they decide to access a clinic. Building on our prior research and collaborations with key community stakeholders providing services to YBMSM and with research experts, we will develop and pilot test "PrEP-Talk," a brief 3-session, 4-week dyad-level intervention, with up to 3 booster sessions on PrEP adherence for any dyad in which the YBMSM index participant (IP) starts PrEP; the IP is the focus of the intervention. IPs randomized to the control will receive regular care. We will accomplish our goal with the following specific aims:

1. To develop and manualize "PrEP-Talk," which aims to increase PrEP uptake and adherence among YBMSM. This will be done through qualitative formative research (3 focus groups with 12-18 YBMSM and CF dyads, N=24-36); partnering with our community advisory board (CAB; comprised of individuals knowledgeable about HIV work with YBMSM); and field tests of the intervention with 5 YBMSM and CF dyads (N=10).
2. Examine feasibility, acceptability and indicators of preliminary efficacy of "PrEP-Talk" on PrEP uptake and adherence among YBMSM. This will be accomplished through a small-scale pilot randomized controlled trial (RCT) with 30 dyads (YBMSM and CFs) in the intervention and 30 dyads in the usual care control arm (N=120). We will conduct assessments of all participants (IPs and CFs) at baseline, 3-months and 6-months post-baseline. We will collect urine samples as a biomarker of PrEP uptake from all YBMSM IPs who report use of PrEP in both arms.

Our intervention may increase PrEP uptake and adherence among YBMSM, thereby helping to reduce HIV incidence and reducing a critical public health disparity. If the proposed intervention shows trends for feasibility, acceptability and indicators of preliminary efficacy for increasing PrEP uptake among YBMSM, we will pursue funding for a full-scale R01-funded RCT.

ELIGIBILITY:
Inclusion Criteria:

age: Index and Close Friends: 18-29 Gender: male assigned at birth or identifies as male or gender queer/non-binary/gender non-conforming; Close Friend none Racial/Ethnic Background: Index: Black/African American or Multiracial and partially identifies as Black/African American' Close Friend: no racial/ethnic restriction Sexual Orientation: Index: self-identify as gay or bisexual; Close Friend: none HIV status: Index must be currently HIV negative; Close Friend: none Currently using PrEP: Index must be not currently using PrEP; Close Friend:none Index must have a close friend with whom they talk regularly about important topics such as sexual health. Close Friend: none.

Close Friend must have a close friend who is Black and gay or bisexual betwen the ages of 18-29.

Close Friend must be willing to support their friend on sexual health goals for HIV prevention.

-

Exclusion Criteria:

Participants are ineligible if they do not meet eligibility requirements stated above.

-

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The index participants must be self-identified as male or male gender expression. Their close friends (whom they choose) may be any gender or gender expression.
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Decision to Begin PrEP | 6 months
  The primary outcome is evidence that the participant has decided to begin PrEP

CONTACTS AND LOCATIONS:
Locations (1):
- Matt Mutchler, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We intend to comply fully with the NIH policy on Data Sharing. Data resulting from the proposed research will be shared with external researchers who request them. Our results will be available to other researchers, public health workers, healthcare professionals, and community leaders who are interested in adherence interventions among PLWHA. Constraints imposed by human research subjects protection regulations (e.g., HIPAA Protected Health Information) and RAND's IRB will be recognized as allowed by NIH. External researchers interested in investigator data, survey instruments, and other research methodology and procedures will obtain this information through collaborative agreements (e.g., data use agreements) with the Principal Investigator and Co-Investigators, as required by NIH's data sharing policy.
Time Frame: We intend to comply fully with the NIH policy on Data Sharing. Data resulting from the proposed research will be shared with external researchers who request them. Our results will be available to other researchers, public health workers, healthcare professionals, and community leaders who are interested in adherence interventions among PLWHA. Constraints imposed by human research subjects protection regulations (e.g., HIPAA Protected Health Information) and RAND's IRB will be recognized as allowed by NIH. External researchers interested in investigator data, survey instruments, and other research methodology and procedures will obtain this information through collaborative agreements (e.g., data use agreements) with the Principal Investigator and Co-Investigators, as required by NIH's data sharing policy.
Access Criteria: We intend to comply fully with the NIH policy on Data Sharing. Data resulting from the proposed research will be shared with external researchers who request them. Our results will be available to other researchers, public health workers, healthcare professionals, and community leaders who are interested in adherence interventions among PLWHA. Constraints imposed by human research subjects protection regulations (e.g., HIPAA Protected Health Information) and RAND's IRB will be recognized as allowed by NIH. External researchers interested in investigator data, survey instruments, and other research methodology and procedures will obtain this information through collaborative agreements (e.g., data use agreements) with the Principal Investigator and Co-Investigators, as required by NIH's data sharing policy.